CLINICAL TRIAL: NCT05028881
Title: Serological Responses to SARS-CoV-2 and Their Temporal Pattern in HIV Infected Persons
Brief Title: COVID-19 Serology in People Living with HIV in Hong Kong
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Shui-Shan Lee, MD, Research Professor, Chinese University of Hong Kong
Other Study IDs: Protocol HIV_COVID-19
Record Dates: First submitted 2021-08-28; First posted 2021-08-31 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-08

CONDITIONS: HIV Infections; SARS-CoV-2 Infection; Vaccination; Infection
Keywords: HIV; COVID-19; SARS-CoV-2 vaccination; co-infection; antibody responses
MeSH Terms: conditions — HIV Infections; COVID-19; Infections; Coinfection | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples would be archived for immunological testing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HIV positive: No interventions
  Interventions: Other: blood sampling
- HIV uninfected: No interventions
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — blood sampling for determining antibody responses

SUMMARY:
Immunodeficiency associated with human immunodeficiency virus (HIV) infection could predispose people living with HIV/AIDS (PLHA) to defective serological responses following infection or vaccination. To evaluate the health outcomes of coronovirus disease-2019 (COVID-19) and HIV co-infection, PLHA and HIV-uninfected persons in Hong Kong are invited to join a study for understanding their clinical characteristics and for tracking their levels of antibodies against severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) over a one-year observation period after infection or vaccination. The results could inform the development of prevention and control strategy for PLHA in response to the emerging coronavirus threats.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the health outcomes of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) co-infection in people living with HIV/AIDS (PLHA) in Hong Kong, with the specific objectives of (a) describing the clinical and immunological characteristics of coronavirus diseases-2019 (COVID-19) in PLHA; (b) tracking the CD (cluster of differentiation) 4/CD8 lymphocytes changes following SARS-CoV-2 infection; (c) assessing the temporal changes of SARS-CoV-2 serology profile of PLHA following SARS-CoV-2 transmission and vaccination.

This is a descriptive study involving the analyses of data derived from the testing of PLHA and non-infected controls at different time-points, following SARS-CoV-2 infection / COVID-19 or vaccination, in conjunction with routinely collected clinical data in the setting of Hong Kong.

The total number of subjects to be recruited is 800, of which 50 would be HIV/SARS-CoV-2 co-infected persons. In order that their serological responses to SARS-CoV-2 could be interpreted in perspective, 400 HIV uninfected adults would be recruited for comparison. Separately, 400 PLHA and 50 healthy adults who have received SARS-CoV-2 vaccination would be recruited to form another control group.

Blood sampling would be performed upon diagnosis of COVID-19 disease when a SARS-CoV-2 infected person is hospitalized for treatment, or after vaccination. This would be repeated after discharge for hospitalized patients and on follow-up at the following time-points: 3, 6, 12, 18 and 24 months. Plasma would be separated from the collected blood samples and stored at -20°C before testing. The levels of antibody to SARS-CoV-2 nucleocapsid and spike protein would be measured using enzyme linked immunosorbent assay (ELISA) method, while surrogate virus neutralization test (sVNT) would be performed to track the changes of sero-protection. .

ELIGIBILITY:
Inclusion Criteria:

* adults of age 18 or above, with
* known HIV status
* infection with SARS-CoV-2 or completion of vaccination against SARS-CoV-2

Exclusion Criteria:

* unable to communicate in written/spoken Chinese or English
* concurrent mental illnesses
* prisoners
* absence of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People living with HIV and HIV uninfected persons who have been diagnosed with SARS-CoV-2 infection or have received vaccination against the virus.
Sampling Method: Non-Probability Sample
Enrollment: 488 (Actual)
Dates: Start 2020-05-16 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 antibody early response to infection | 3 months
  proportion antibody positive within 3 months of infection
SARS-CoV-2 antibody early response to vaccination | 3 months
  proportion antibody positive within 3 months of vaccination

SECONDARY OUTCOMES:
SARS-CoV-2 sustained post-infection antibody response | 1 year
  proportion antibody positive at one year after infection
SARS-CoV-2 sustained vaccination response | 1 year
  proportion antibody positive at one year after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Shui Shan Lee, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Shui Shan Lee, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No
Individual data are kept in confidence and would not be available to researchers outside the study, as has been bound by ethics approval